CLINICAL TRIAL: NCT02410759
Title: Carbetocin Versus Oxytocin in the Management of Atonic Post Partum Haemorrhage (PPH) in Women Delivered Vaginally: A Randomised Controlled Trial
Brief Title: Carbetocin Versus Ergometrine in the Management of Atonic Post Partum Haemorrhage (PPH) in Women Delivered Vaginally
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPH5
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Ergonovine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbetocin (Active Comparator): 100 women with atonic PPH will receive Carbetocin 100 µgm slowly IM
  Interventions: Drug: Carbetocin
- Ergometrine (Active Comparator): 100 women with atonic PPH will receive Ergometrine 0.5mg IM
  Interventions: Drug: Ergometrine

INTERVENTIONS:
Drug: Carbetocin — 100 women with atonic PPH will receive Carbetocin 100 µgm IM
  Arms: Carbetocin
Drug: Ergometrine — 100 women with atonic PPH will receive Ergometrine 0.5 µgm IM
  Arms: Ergometrine

SUMMARY:
200 women will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive ergometrine 0.5mg (methergin®, Novartis, Switzerland).

DETAILED DESCRIPTION:
Obstetric haemorrhage remains one of the major causes of maternal death in both developed and developing countries. Postpartum haemorrhage (PPH) is defined as a blood loss >500 ml more of blood from the genital tract within 24 hours of the birth of a baby. PPH can be minor (500-1000 ml) or major (more than 1000 ml). The most frequent cause of PPH is uterine atony, contributing up to 80 % of the PPH cases.

Risk factors of atonic PPH include multiple pregnancy, placenta previa, previous PPH, body mass index (BMI) >30, prolonged labour, fetal macrosomia>4kg and primipara> 40 years.

Oxytocin is currently the uterotonic of first choice. It has proven to decrease the incidence of PPH by 40 % and has a rapid onset of action and a good safety profile. A disadvantage of oxytocin is its short half-life of 4-10 min, regularly requiring a continuous intravenous infusion or repeated intramuscular injections.

Carbetocin is a long-acting oxytocin analogue indicated for the prevention of uterine atony after child birth by cesarean section (CS) under epidural or spinal anaesthesia. Carbetocin has a rapid onset of action (within 1-2 min) and a prolonged duration of action (approximately 1 h) because of sustained uterine response with contractions of higher amplitude and frequency. Its safety profile is comparable to that of oxytocin The study will be conducted in Cairo university hospitals and BeniSuef university hospitals. All patients attending the labour ward will be invited to participate in the study in case they develop PPH, the invitation will include a clear full explanation of the study. Only patients signing informed written consents will participate in the study. All women will receive a prophylactic dose of oxytocin 5 i.u after delivery of the anterior shoulder.

200 women with atonic PPH will be randomly divided into 2 equal groups using computer generated random numbers. Group 1 will receive Carbetocin 100 µgm (Pabal® Ferring, UK) and group 2 will receive ergometrine 0.5mg (Methergine®, Novartis, Switzerland). The investigators will not include a control group for ethical reasons.

Once atonic PPH is diagnosed, 2 14-gauge cannulas will be inserted and a crystalloid intravenous (iv) infusion will be started. The allocated drug will be diluted in 10ml saline and will be given slowly iv, the fundus will be rubbed, A Foley's catheter will be inserted and a fluid balance chart will be commenced, pulse and blood pressure will be recorded every 15 minutes, venepuncture will be done for cross matching 4 units of blood, full blood count and coagulation screen.

The uterine tone and amount of bleeding will be noted and the need for further uterotonic agents will be determined 2 minutes after giving the drug. Blood loss will be estimated through weighing the swabs and using pictorial charts. Blood haemoglobin will be assessed 24 hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Women with atonic PPH.

Exclusion Criteria:

* Gestational age <37 weeks.
* Hypertension.
* Preeclampsia.
* Cardiac, renal or liver diseases
* Epilepsy.
* Known hypersensitivity to Carbetocin

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Need for other uterotonics | 2 minutes after giving the drug.
  The uterus will be felt for the tone.

SECONDARY OUTCOMES:
Development of major PPH | 10 minutes after giving the drug
  Swabs will be weighed and pictorial charts will be used to estimate the bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany M Hassan, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - BeniSuef University hospitals, BeniSuef
  - Cairo university hospitals, Cairo

REFERENCES:
- [Background] Moertl MG, Friedrich S, Kraschl J, Wadsack C, Lang U, Schlembach D. Haemodynamic effects of carbetocin and oxytocin given as intravenous bolus on women undergoing caesarean delivery: a randomised trial. BJOG. 2011 Oct;118(11):1349-56. doi: 10.1111/j.1471-0528.2011.03022.x. Epub 2011 Jun 14. PMID 21668768
- [Background] Winter C, Macfarlane A, Deneux-Tharaux C, Zhang WH, Alexander S, Brocklehurst P, Bouvier-Colle MH, Prendiville W, Cararach V, van Roosmalen J, Berbik I, Klein M, Ayres-de-Campos D, Erkkola R, Chiechi LM, Langhoff-Roos J, Stray-Pedersen B, Troeger C. Variations in policies for management of the third stage of labour and the immediate management of postpartum haemorrhage in Europe. BJOG. 2007 Jul;114(7):845-54. doi: 10.1111/j.1471-0528.2007.01377.x. PMID 17567419
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518